CLINICAL TRIAL: NCT01319162
Title: To Estimate the Prevalence of PCOS in Obese Premenopausal Women and Elucidate How They Respond to a Weight Reduction Treatment Program
Brief Title: Prevalence of Polycystic Ovary Syndrome (PCOS) in Obese Premenopausal Women
Status: Completed | Type: Observational
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Other Study IDs: Prevalence-PCOS-Obesity
Record Dates: First submitted 2011-03-18; First posted 2011-03-21 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Women with PCOS: All obese women between 18 and 50 years diagnosed with PCOS referred to a weight reduction treatment program at the Sahlgrenska Obesity Center at Sahlgrenska University hospital
  Interventions: Other: Weight reduction regimen
- Women without PCOS: All obese women between 18 and 50 years not diagnosed with PCOS referred to a weight reduction treatment program at the Sahlgrenska Obesity Center at Sahlgrenska University hospital
  Interventions: Other: Weight reduction regimen

INTERVENTIONS:
Other: Weight reduction regimen — The dietary intervention begins with a 12-weeks VLCD/LCD period. The diet comprise of 3 to 5 portions liquid diet with a daily energy intake of 450-800 kcal. In addition, patients will be encouraged to drink 1,5-2L daily of non-caloric beverages (<6 kcal/100 ml). All patients will have scheduled nurse visits at week 0 (baseline), 2, 5, 8, and 12. At these visits general well-being and body weight will be monitored. The patient will also be given support and counselling to enhance compliance to the VLCD/LCD diet.

SUMMARY:
Between 40% and 85% of women with Polycystic Ovary Syndrome (PCOS) are overweight or obese and obesity is closely linked to the development of PCOS. Although it is well established that obesity increases the severity of the clinical features of PCOS, data regarding the prevalence of PCOS in obese women and the change in body weight in women with PCOS over time are scares. In a prevalence study it was investigated whether obesity increases the risk of PCOS in the general population and they demonstrated that the prevalence rate of PCOS in underweight, normal-weight, overweight, and obese women were 8.2, 9.8, 9.9, and 9.0%, respectively, similar to that observed in the general population. These results suggest that the risk of PCOS is only minimally increased with obesity. On the other hand, in a Spanish prevalence study among overweight and obese subjects, they demonstrated a 28.3% prevalence of PCOS, which is markedly higher compared with the 5.5% prevalence of PCOS in lean women in Spain.

First the investigators aim to estimate the prevalence/probability of PCOS among obese, premenopausal women (between 18 and 50 years) with no symptoms of classic menopausal symptoms in Sweden. Secondly, to elucidate whether women diagnosed with PCOS respond to standard weight reduction regime to the same extent as women without PCOS.

ELIGIBILITY:
Inclusion Criteria:

PCOS diagnostic criteria should be the presence of both clinical and/or biochemical hyperandrogenism and/or oligo-/amenorrhea and/or polycystic ovaries (PCO).

Exclusion Criteria:

1. Exclusion of other endocrine disorders such as hyperprolactinemia (s-prolactin < 27µg/L), nonclassic congenital adrenal hyperplasia (17-hydroxyprogesterone < 3nmol/L), and androgen secreting tumors.
2. Pregnancy or breastfeeding the last 6 months.
3. Any sign of climacteric symptoms.
4. Language barrier or disabled person with reduced ability to understand information.
5. Oral contraceptives and insulin sensitizing agents is commonly used among women with PCOS since it may interfere with hormone profile. As the prevalence of PCOS can be assumed to be increased among women using oral contraceptives and insulin sensitizing agents, they are included but analyzed separately.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All obese women between 18 and 50 years referred to a weight reduction treatment program at the Sahlgrenska Obesity Center at Sahlgrenska University hospital will, after oral and written informed consent, be screened for the diagnosis of PCOS according to NIH or Rotterdam diagnostic criteria depending on the availability of ultrasonography.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2011-03-30 (Actual); Primary Completion 2017-01-11 (Actual); Study Completion 2017-01-11 (Actual)

PRIMARY OUTCOMES:
Prevalence/probability of PCOS among obese, premenopausal women (between 18 and 50 years) with no symptoms of classic menopausal symptoms in Sweden. | Within one month after first visit
  Screening for PCOS among obese women includes menstrual history, clinical and biochemical signs of hyperandrogenism and polycystic ovaries on ultrasound measure in women with one of signs included in the diagnosis of the syndrome.

SECONDARY OUTCOMES:
Response to weight reduction regime among obese women with and without PCOS | One year after inclusion
Food frequency | Within one month after measure
Health Related Quality of Life | Screening and one year later
Symptoms of anxiety and depression | Screening and after one year
Changes in sex steroids and other related hormones | Screening and after 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska Obesity Center at Sahlgrenska University hospital, Gothenburg, Sweden

REFERENCES:
- [Derived] Kataoka J, Olsson M, Lindgren E, Larsson I, Schmidt J, Benrick A, Stener-Victorin E. Effects of weight loss intervention on anxiety, depression and quality of life in women with severe obesity and polycystic ovary syndrome. Sci Rep. 2024 Jun 12;14(1):13495. doi: 10.1038/s41598-024-63166-w. PMID 38866860
- [Derived] Kataoka J, Stener-Victorin E, Schmidt J, Larsson I. A prospective 12-month structured weight loss intervention in women with severe obesity and polycystic ovary syndrome: Impact of weight loss on eating behaviors. Acta Obstet Gynecol Scand. 2024 Aug;103(8):1615-1624. doi: 10.1111/aogs.14867. Epub 2024 May 8. PMID 38717931
- [Derived] Kataoka J, Larsson I, Lindgren E, Kindstrand LO, Schmidt J, Stener-Victorin E. Circulating Anti-Mullerian hormone in a cohort-study of women with severe obesity with and without polycystic ovary syndrome and the effect of a one-year weight loss intervention. Reprod Biol Endocrinol. 2022 Oct 29;20(1):153. doi: 10.1186/s12958-022-01022-0. PMID 36309748
- [Derived] Kataoka J, Larsson I, Bjorkman S, Eliasson B, Schmidt J, Stener-Victorin E. Prevalence of polycystic ovary syndrome in women with severe obesity - Effects of a structured weight loss programme. Clin Endocrinol (Oxf). 2019 Dec;91(6):750-758. doi: 10.1111/cen.14098. Epub 2019 Oct 1. PMID 31529511